CLINICAL TRIAL: NCT05411653
Title: Combined Effects of Xbox Kinect Virtual Reality and Motor Imagery on Lower Limb Function, Dynamic Balance and Gait in Chronic Stroke Patients
Brief Title: Xbox Kinect Virtual Reality and Motor Imagery on Lower Limb Function in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0213
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality training with motor imagery (Experimental): Xbox Kinect VR with MI training Five Xbox Kinect gaming will be selected and explained to the patients for the virtual training session
  Interventions: Other: Virtual reality training with motor imagery
- Conventional physical therapy (Active Comparator): a range of motion exercises, muscle strengthening, functional training, balance training, and gait training. T
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Virtual reality training with motor imagery — comprised of 30 minutes, VRT (15 minutes) and MI (15 minutes) daily for 3 days respectively. Five Xbox Kinect gaming will be selected and explained to the patients for the virtual training session and additional 15 minutes will be given to them for practice. The games consists of 20,000 water leaks, river rush, reflex ridge, soccer and football for the patients.
  Arms: Virtual reality training with motor imagery
Other: Conventional physical therapy — range of motion exercises, muscle strengthening, functional training, balance training, and gait training. The specific tasks will be selected by the therapist based on the requirement of each patient. It will be performed for 30 minutes for 3 days a week for 6 weeks
  Arms: Conventional physical therapy

SUMMARY:
As virtual reality has therapeutic benefits and improves motor learning by practicing exercises in environment that analogue and mimic occasions and events of real world, as VR is designed and tailored according to the need of patient so it may address the individual issues whereas motor imagery uses explicit learning process for muscle activation and movement. Therefore their combination may yield better outcomes in terms of lower limb function and dynamic mobility, so there is a need to assess the combined effects of Xbox kinect gaming with motor imagery in chronic stroke patients.

DETAILED DESCRIPTION:
Stroke is focal neurological disorder that occurs due to the compromised blood flow to the brain. It results in mobility deficit, functional and gait impairment. Multiple rehabilitation methods have been designed and used, motor imagery (MI) and virtual reality (VR) are among the emerging techniques that are being used for the rehabilitation of patients with neurological conditions that improve motor learning through explicit and implicit processes.

After stroke the residual symptoms such as muscle hyper tonicity, attention deficiency, hemi neglect, abnormal reflexes and sensorimotor functional impairment may persist. Additional to these neurological symptoms certain balance issues may cause decrease in proprioception, muscle strength, increased load on non-paretic extremity and postural oscillations. It has been reported that every year approximately 25.7 million people survive stroke attacks, 6.5 million die because of stroke and 113 million people have disability-adjusted life-years.

Kinect based rehabilitation and virtual feedback have shown relevant activation changes in the primary sensorimotor cortex and can be responsible for that part of brain reorganization for improving in upper limb in stroke patients. Use of exer gaming is one of the emerging technologies that are being used for the physical, cognitive and motor rehabilitation of stroke patients. It is combination of video games and motion sensors incorporated in a virtual reality environment that engage the patients and improves motor learning therefore activating the motor areas of the brain for long term results.

Non immersive virtual reality gaming has been used for improving balance among the stroke patients. Not only is it considered more beneficial as compared to the conventional therapies but also maintains the interest of patients in their rehabilitation protocol. The Kinect based games use sensors that catch movements of the patients and they are able to watch them in real time with immediate feedback that becomes a source of motivation for them.

Xbox Kinect virtual gaming creates 3D environment with sensors and requires no controllers for patients to perform exercise whereas motor imagery is a state in which a particular motor action is internally activated without any motor output. Not only is VR and MI training motivating as compare to conventional therapies but also provide positive learning experience and neuroplasticity. With xbox kinect based VR therapies and MI, the exercise plan is tailored according to the needs of the patient.

It will be a single blinded randomized control trial in which control group will be given conventional physiotherapy protocol for 30 minutes and experimental group will receive the VR and MI training with conventional treatment for a total 60 minutes, 3 days a week for 6 weeks. Motor function will be assessed by fugl-meyer scale (LE), dynamic mobility by berg balance scale and 6 minute walk test, quality of life by barthel index and gait with dynamic gait index. Patient will be assessed at baseline and at the end of six weeks. The data will be analyzed using SPSS 25 software.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are 45-65 years of age
* Participants who have had their first stroke attack at least 6 months prior
* A score of 21 or greater on the Mini-Mental State Examination (MMSE)
* Participants who were not diagnosed with visual or auditory issues
* Volunteers should be able to walk at least 10 meters with or without assistive devices
* The patient shouldn't be taking any medicine that can have an impact on the gait or balance.

Exclusion Criteria:

* Patients younger than 45 years of age.

  * Patients suffering from any condition that requires medical attention such as uncontrolled blood pressure or angina.
  * Musculoskeletal impairments of the lower extremity.
  * Patients with psychological or neurological problems other than stroke

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index DGI | 6th week
  Clinical tool to assess gait, balance and fall risk. It evaluates not only usual steady-state walking, but also walking during more challenging tasks
Berg Balance Scale BBS | 6th week
  Objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks.
Fugl-Meyer Scale for lower extremity | 6th week
  This clinical tool is for assessment of lower limb function. It is a reliable and valid tool. Interrater and intrarater reliability coefficients are reported to be >0.85 for both upper and lower limb) the domain subscales and the entire scale.
Six Minute Walk Test | 6th week
  It is used to assess aerobic capacity and endurance.

SECONDARY OUTCOMES:
Barthel index | 6th week
  It is functional independence measure.

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee HC, Huang CL, Ho SH, Sung WH. The Effect of a Virtual Reality Game Intervention on Balance for Patients with Stroke: A Randomized Controlled Trial. Games Health J. 2017 Oct;6(5):303-311. doi: 10.1089/g4h.2016.0109. Epub 2017 Aug 3. PMID 28771379
- [Background] Aslam M, Ain QU, Fayyaz P, Malik AN. Exer-gaming reduces fall risk and improves mobility after stroke. J Pak Med Assoc. 2021 Jun;71(6):1673-1675. doi: 10.47391/JPMA.875. PMID 34111095
- [Background] Bao X, Mao Y, Lin Q, Qiu Y, Chen S, Li L, Cates RS, Zhou S, Huang D. Mechanism of Kinect-based virtual reality training for motor functional recovery of upper limbs after subacute stroke. Neural Regen Res. 2013 Nov 5;8(31):2904-13. doi: 10.3969/j.issn.1673-5374.2013.31.003. PMID 25206611
- [Background] Silva S, Borges LR, Santiago L, Lucena L, Lindquist AR, Ribeiro T. Motor imagery for gait rehabilitation after stroke. Cochrane Database Syst Rev. 2020 Sep 24;9(9):CD013019. doi: 10.1002/14651858.CD013019.pub2. PMID 32970328
- [Background] Bovonsunthonchai S, Aung N, Hiengkaew V, Tretriluxana J. A randomized controlled trial of motor imagery combined with structured progressive circuit class therapy on gait in stroke survivors. Sci Rep. 2020 Apr 24;10(1):6945. doi: 10.1038/s41598-020-63914-8. PMID 32332810
- [Background] Lin RC, Chiang SL, Heitkemper MM, Weng SM, Lin CF, Yang FC, Lin CH. Effectiveness of Early Rehabilitation Combined With Virtual Reality Training on Muscle Strength, Mood State, and Functional Status in Patients With Acute Stroke: A Randomized Controlled Trial. Worldviews Evid Based Nurs. 2020 Apr;17(2):158-167. doi: 10.1111/wvn.12429. Epub 2020 Mar 25. PMID 32212254
- [Background] Askin A, Atar E, Kocyigit H, Tosun A. Effects of Kinect-based virtual reality game training on upper extremity motor recovery in chronic stroke. Somatosens Mot Res. 2018 Mar;35(1):25-32. doi: 10.1080/08990220.2018.1444599. Epub 2018 Mar 13. PMID 29529919
- [Background] Malik AN, Masood T. Effects of virtual reality training on mobility and physical function in stroke. J Pak Med Assoc. 2017 Oct;67(10):1618-1620. PMID 28955088
- [Background] Chanpimol S, Seamon B, Hernandez H, Harris-Love M, Blackman MR. Using Xbox kinect motion capture technology to improve clinical rehabilitation outcomes for balance and cardiovascular health in an individual with chronic TBI. Arch Physiother. 2017;7:6. doi: 10.1186/s40945-017-0033-9. Epub 2017 May 31. PMID 28824816
- [Background] In T, Lee K, Song C. Virtual Reality Reflection Therapy Improves Balance and Gait in Patients with Chronic Stroke: Randomized Controlled Trials. Med Sci Monit. 2016 Oct 28;22:4046-4053. doi: 10.12659/msm.898157. PMID 27791207
- [Background] Im H, Ku J, Kim HJ, Kang YJ. Virtual Reality-Guided Motor Imagery Increases Corticomotor Excitability in Healthy Volunteers and Stroke Patients. Ann Rehabil Med. 2016 Jun;40(3):420-31. doi: 10.5535/arm.2016.40.3.420. Epub 2016 Jun 29. PMID 27446778
- [Background] Gibbons EM, Thomson AN, de Noronha M, Joseph S. Are virtual reality technologies effective in improving lower limb outcomes for patients following stroke - a systematic review with meta-analysis. Top Stroke Rehabil. 2016 Dec;23(6):440-457. doi: 10.1080/10749357.2016.1183349. Epub 2016 May 30. PMID 27237336
- [Background] Bae YH, Ko Y, Ha H, Ahn SY, Lee W, Lee SM. An efficacy study on improving balance and gait in subacute stroke patients by balance training with additional motor imagery: a pilot study. J Phys Ther Sci. 2015 Oct;27(10):3245-8. doi: 10.1589/jpts.27.3245. Epub 2015 Oct 30. PMID 26644684
- [Background] Park DS, Lee DG, Lee K, Lee G. Effects of Virtual Reality Training using Xbox Kinect on Motor Function in Stroke Survivors: A Preliminary Study. J Stroke Cerebrovasc Dis. 2017 Oct;26(10):2313-2319. doi: 10.1016/j.jstrokecerebrovasdis.2017.05.019. Epub 2017 Jun 9. PMID 28606661